CLINICAL TRIAL: NCT05176457
Title: A Communication Tool's Evaluation on Intensive Care Patients Equipped With Ventilation Systems.
Brief Title: Communication Tool Evaluation on Intensive Care Patients.
Acronym: PICT'REA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0427
Record Dates: First submitted 2021-10-21; First posted 2022-01-04 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Communication, Nonverbal
Keywords: intensive care; communication tool; invasive ventilation; speaking impairment; technology
MeSH Terms: conditions — Nonverbal Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEFORE PICT'REA introduction (No Intervention): Patients will have the usual communication tools (pen and paper, hands gestures...)
- AFTER PICT'REA introduction (Experimental): Patients will be given a tablet to communicate with the caregivers whenever needed
  Interventions: Other: communication tool PICT'REA

INTERVENTIONS:
Other: communication tool PICT'REA — The pictograms communication tool "PICT'REA" will be available to patients with invasive ventilation systems preventing them from speaking
  Arms: AFTER PICT'REA introduction

SUMMARY:
The present study evaluate the impact of a communication tool "PICT'REA" on patients in reanimation units, equipped with ventilation systems, preventing them from speaking.

The app consists of simple pictograms allowing simple communication between patients and the reanimation care team.

The study will assess the quality of communication before and after the introduction of the communication tool in the reanimation unit.

DETAILED DESCRIPTION:
Invasive mechanical ventilation is commonly used in intensive care, in sedated patients but also in perfectly conscious patients, and this on a daily basis.

For these patients, the resulting deprivation of oral expression is a major source of stress and discomfort. On the side of the caregivers, the difficulty of comprehension is a source of frustration on a daily basis.

Thus PICT'REA has been developped in order to help patients and caregivers to better understand each other during invasive ventilation.

PICT'REA is a tool in the form of a mobile app with simple pictograms allowing simple communication (Yes/No/Pain chart...).

The study will analyze the quality of communication between patients and caregivers before and after the introduction of the application:

* Before setting up the tool: control group

  * Over a period of 6 months
  * In the multi-purpose resuscitations of Cardio Vascular Surgery and Neurosurgery.
* After setting up the tool:

  * Over a period of 6 months
  * In the same departments.

The analyses consists of various questionnaires :

* the modified Ease of Communication Scale,
* a Short questionnaire in 3 questions for caregivers,
* IPREA questionnaire for patients,
* Evaluation of the usability of the system by System Usability Scale questionnaire,
* Evaluation of the attractiveness of the system by Attrackdiff questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in intensive care or intensive care
* ventilated on a tracheostomy or an orotracheal intubation tube for> 24 hours
* not too agitated or too sedated (RASS -1 to +2) for> 24 hours
* Confusion Assessment Method (CAM) ICU negative
* Speak or read French

Exclusion Criteria:

Inability to use the device:

* Blind or visually impaired
* Severe paresis of the upper limbs
* No understanding of the tool.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Ease of Communication | before PICT'REA introduction (Baseline)
  The modified Ease of Communication Scale (ECS), comprising 8 questions of 1 to 5 points, for a maximum total of 40 points. The lower the score, the easiest the communication is.
  This is regarding patients using traditional communication methods (slate, alphabet, lip reading, etc.)
Ease of Communication | after PICT'REA introduction (6 months)
  The modified Ease of Communication Scale (ECS), comprising 8 questions of 1 to 5 points, for a maximum total of 40 points. The lower the score, the easiest the communication is.
  This is regarding patients using the PICT REA application.

CONTACTS AND LOCATIONS:
Overall Officials: Fanny VARDON-BOUNES, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France